CLINICAL TRIAL: NCT00294736
Title: A Two-Stage Phase 1 Dose Escalation Pharmacokinetic Study of Tarceva® (Erlotinib) in Patients With Stage IIIB/IV Non-small Cell Lung Cancer Who Continue To Smoke After Failure of One or Two Prior Chemotherapy Regimens
Brief Title: A Two-Stage Phase 1 Dose Escalation Pharmacokinetic Study of Tarceva in Patients With Stage IIIB/IV Non-small Cell Lung Cancer Who Continue to Smoke After Failure of One or Two Prior Chemotherapy Regimens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSI-774-107; 2005-003883-46 (EudraCT Number)
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: NSCLC
Keywords: lung cancer; erlotinib; NSCLC; smokers
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Arm A (Tarceva MTD established in Part I)
  Interventions: Drug: Tarceva
- Arm B (Experimental): Arm B (150 mg Tarceva daily).
  Interventions: Drug: Tarceva

INTERVENTIONS:
Drug: Tarceva — Dose Escalation: 150-350+ mg/day

SUMMARY:
This is a multicenter, open-label, randomized phase 1 study of escalating doses of Tarceva in patients with advanced NSCLC who currently smoke.

Part I will establish the maximum tolerated dose (MTD) of Tarceva in current smokers.

In Part II, patients will be randomized 1:1 to two treatment groups: Arm A (Tarceva MTD established in Part I) and Arm B (150 mg Tarceva daily). Patients in both arms will be treated for two weeks and then have pharmacokinetic samples collected on day 14. Part II is open as of Nov-2006.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IIIB/IV NSCLC;
* Must have received 1 or 2 prior chemotherapy regimens for advanced NSCLC and now have progressive disease;
* Must have recovered from any treatment-related toxicities prior to registration, except for alopecia, grade 1 fatigue, or grade 1 neurotoxicity;
* A current cigarette smoker (minimum of 10 cigarettes per day for >= 1 year and have a positive test for cotinine) despite advice and support to quit;
* Age >= 18 years;
* ECOG PS 0-1 and predicted life expectancy >= 12 weeks;
* Previous surgery is permitted provided that wound healing has occurred prior to registration;
* Adequate hematopoietic, hepatic and renal function defined as follows: ANC >= 1.5 x 10^9/L, platelets >= 100 x 10^9/L, bilirubin <= 1.5 x ULN, ALT <= 2.5 x ULN (or 5 x ULN in case of liver metastases), creatinine <= 1.5 x ULN;
* No prior treatment with Tarceva or gefitinib (or other drug with significant activity against EGFR (eg, cetuximab and/or ZD6474));
* Patients with reproductive potential must practice effective contraceptive measures throughout the study. Women of child-bearing potential must provide a negative pregnancy test within 14 days prior to registration;
* Accessible for repeat dosing and follow-up.

Exclusion Criteria:

* Any concurrent anticancer cytostatic or cytotoxic chemotherapy;
* Concomitant CYP3A4 or CYP1A2 inducers/inhibitors (or during 14 days prior to study) with the exception of tobacco;
* Other active malignancies, unless disease-free and without cancer-specific therapy for at least the last 5 years. Basal or squamous cell skin cancers are not excluded;
* Significant history of cardiac disease unless the disease is well-controlled;
* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with the patient's ongoing participation in the study;
* History of any psychiatric condition that might impair the patient's ability to understand or comply with the requirements; of the study or to provide informed consent.
* Gastrointestinal abnormalities, including inability to take oral medication, requirement for IV alimentation, active peptic ulcer or prior surgical procedures affecting absorption;
* Clinically significant ophthalmologic abnormalities;
* Pregnant or breast-feeding females. Males or females not practicing effective birth control;
* Symptomatic brain metastases which are not stable, require steroids, or that have required radiation within the last 28 days;
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drug;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To establish the MTD of Tarceva in currently smoking patients with stage IIIB/IV NSCLC. | 2 years

SECONDARY OUTCOMES:
To evaluate the survival of currently smoking patients with stage IIIB/IV NSCLC when given Tarceva at the MTD and 150 mg. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — OSI Pharmaceuticals
Locations (9):
- United States (2):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
- United Kingdom (7):
  - University of Edinburgh,Division of Oncology,, Edinburgh, Scotland
  - Aberdeen Royal Infirmary, Aberdeen
  - Ninewells Hospital, Dundee
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Sir Bobby Robson Cancer Trials Research Centre, Newcastle upon Tyne
  - Department of Oncology, Sheffield
  - Royal Marsden Hospital, Sutton